CLINICAL TRIAL: NCT06002256
Title: Mostafa Maged Maneuver in Comparison With Bimanual Uterine Compression to Control Post-partum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mostafa Maged Ali, principal investigator, Ministry of Health and Population, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (598 ) , Al-Azhar university
Record Dates: First submitted 2023-08-06; First posted 2023-08-21 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Post-partum Hemorrhage
Keywords: Mostafa Maged maneuver; Bimanual uterine compression; vaginal delivery; postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : Mostafa Maged maneuver (Active Comparator): The first step in the Mostafa Maged maneuveur step is placing the right hand to the posterior fornix of vaginal canal trying to put pressure on the cervix and the lower part of uterus compressing the anterior and posterior walls of the lower uterine segment. The second point is placing the left hand over the fundus of the uterus and the posterior wall of the uterus from the abdominal part of the pregnant mother (the side of the abdominal skin). The third step is trying to grasp the whole uterus by the two hands abdominally and vaginally against the symphysis pubis as if the uterus is containing or surrounding the symphysis pubis bone, and in this way, getting the anterior and posterior walls of the uterus against each other (compression achieved)
  Interventions: Procedure: Mostafa Maged maneuver
- Group 2 : bimanual uterine compression (Other): Both maneuver s are performed immediately after the delivery of the placenta and foetus, with no uterotonics administered at the onset of these maneuver s. In the event of atony after hand release due to fatigue, 5 IU of oxytocin is administered intravenously as uterotonics.
  the clinician places one hand on the abdomen and the other hand inside the vagina then compresses the uterus between the two hands.
  Interventions: Procedure: Bimanual uterine compression

INTERVENTIONS:
Procedure: Mostafa Maged maneuver — While the patient is on the lithotomy position , The first step in the Mostafa Maged maneuveur step is placing the right hand to the posterior fornix of vaginal canal trying to put pressure on the cervix and the lower part of uterus compressing the anterior and posterior walls of the lower uterine segment. The second point is placing the left hand over the fundus of the uterus and the posterior wall of the uterus from the abdominal part of the pregnant mother (the side of the abdominal skin). The third step is trying to grasp the whole uterus by the two hands abdominally and vaginally against the symphysis pubis as if the uterus is containing or surrounding the symphysis pubis bone, and in this way, getting the anterior and posterior walls of the uterus against each other (compression achieved)
  Arms: Group 1 : Mostafa Maged maneuver
Procedure: Bimanual uterine compression — the clinician places one hand on the abdomen and the other hand inside the vagina then compresses the uterus between the two hands.
  Arms: Group 2 : bimanual uterine compression

SUMMARY:
The current study aimed to investigate the effectiveness of the Mostafa Maged maneuver compared to Bimanual uterine compression in controlling postpartum hemorrhage during vaginal delivery.

The study subjects were categorized into two groups. The first group was managed by the Mostafa Maged maneuver , whereas the second group was managed by routine bimanual uterine compression.

investigators attempted to determine the duration of each maneuver required until the investigator became exhausted, as well as whether or not oxytocin was administered later in each maneuver .

ELIGIBILITY:
Inclusion Criteria:

- female and pregnant

Exclusion Criteria:

* hematological diseases morbid obese smoking

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female pregnant
Enrollment: 200 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Good hemostasis and achieving the uterus contracted | first 3 hours
  no post-partum hemorrhage , we assess this by the amount of bleeding going down and by the atonic status of the uterus at that time
obstetrician does not feel fatigued | during applying the maneuver
  no exhaustion for the obstetrician , and this outcome is told by the investigators themselves

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum general hospital and al azhar university, Cairo, Cairo and Fayoum, Egypt

IPD SHARING:
Plan to Share IPD: No